<<ENTER NHS TRUST LOGO>>





## ChemoBrain Prehab Project: Improving Brain Health After Chemotherapy Through Prehabilitation

| IRAS ID | : 356825 | |
|---|---|---|
| Centre N | lumber: | |
| Study N | umber: | |
| Participa | ant Identification Number for this trial: | |
| CONSENT FORM | | |
| Title of F | Project: ChemoBrain Prehab Project: Improving Brain Health After Chemotherapy Through | n Prehabilitation |
| Name of | Researcher: Katie Hoad, Lancaster University | |
| | | Please Initial Box |
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that any data collected up to the point of my withdrawal may still be used in the study. | |
| 4. | I understand that Lancaster University as the sponsor or regulatory authorities may be granted access to the study records and data for monitoring and auditing purposes. I give permission for these individuals to have access to my records. | |
| 5. | I consent to anonymised information being used in reports, conferences and training events. | |
| 6. | I consent to provide blood samples as per the study schedule. I understand these will be stored securely until the study ends, at which point the samples will be analysed. | |
| 7. | I agree to my direct care team and general practitioner being informed of my participant in the study if any concerns may arise during testing that they should be made aware of. | |
| 8. | I have the option to join the online Microsoft Teams group used in this study. If I decide to join, I agree that my name and email address will be visible to the other members of the group. I understand that all members will be instructed to keep this information confidential and not use it for any purpose outside the study. <i>(optional)</i> | |
| 9. | I confirm that I have had the opportunity to ask any questions and to have them answered. | |
| 10. | I agree to take part in the above study. | |

IRAS ID: 356825

## <<ENTER NHS TRUST LOGO>>





| Name of Participant | Date | Signature |
|-------------------------------|------|-----------|
| Name of Person Taking Consent | Date | Signature |

One copy to be retained by the participant, and one copy to be retained by the research team.